CLINICAL TRIAL: NCT03813459
Title: Subsyndromal Delirium in Intensive Care Unit, a Multicenter Study
Brief Title: Subsyndromal Delirium in Intensive Care Unit
Acronym: SubSynD
Status: Completed | Type: Observational
Sponsor: Centro Hospitalar Lisboa Ocidental (Other Government)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Maria Carolina Vieira Júlio Paulino, Principal Investigator, Centro Hospitalar Lisboa Ocidental
Other Study IDs: UCIP1
Record Dates: First submitted 2019-01-13; First posted 2019-01-23 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Delirium
Keywords: Delirium; Subsyndromal delirium; Intensive Care Unit
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subsyndromal delirium positive: Presence of Subsyndromal delirium in Intensive Care patients
- Delirium positive: Presence of Delirium in Intensive Care patients
- No delirium: Non subsyndromal delirium or delirium in Intensive Care patients

SUMMARY:
Subsyndromal delirium (SSD) is a condition characterized by a less severe cognitive impairment in comparison to delirium. To date there is no published consensus on SSD definitions and has been commonly reported as an intermediate stage between delirium and normal mental states.

SSD encompasses some of the delirium symptoms, and has been diagnosed with Intensive Care Delirium Screening Checklist scale (ICDSC) and Confusion Assessment Method-ICU (CAM-ICU).

The objective of this study is to identify subsyndromal delirium prevalence, the association between SSD and clinical outcomes and understanding the relationship between SSD and conversion to delirium.

The relevance of this study is understanding of subsyndromal delirium in ICU, namely the importance of early presentations of acute brain dysfunction in the patients outcome.

DETAILED DESCRIPTION:
SubSynD is a prospective, observational, multicenter clinical study, involving 400 patients in Intensive Care Units, to assess subsyndromal delirium.

A systematic screening for delirium and subsyndromal delirium (SSD) is done with Intensive Care Delirium Screening Checklist (ICDSC) and Confusion Assessment Method-ICU (CAM-ICU). Scales are applied once per day until ICU discharge or for up to 14 days of being in ICU.

The investigators access three different groups of patients: non-delirium, delirium and subsyndromal delirium. It is intended that either ICDSC or CAM-ICU, paired with a Richmond Agitation and Sedation Scale (RASS) be administered once per day (i.e. with first assessment in the morning). All patients with abnormal CAM-ICU or ICDSC features, beside the underlying cause of delirium and SSD are included. In addition, data regarding baseline demographic and clinical characteristics will be collected as well as data regarding the procedure performed (see Case Report Form (CRF)).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Admission in Intensive care Unit

Exclusion Criteria:

1. Primary neurological diagnosis, with Glasgow Coma Scale (GCS) <14 on ICU admission or in previous days;
2. Blindness or deafness;
3. Aphasia;
4. Inability to communicate in the native language of the country where the study is enrolled;
5. Death during the first 24 hours;
6. Limitation of therapeutic efforts in the Intensive Care Unit admission;
7. Refusal to participate;
8. Previous diagnosis of dementia or psychiatric illness;
9. Readmission in ICU;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with conversion from subsyndromal delirium to delirium during the period of study | 14 days
  ICDSC performed 1 time per day and determine how subsyndromal delirium (ICDSC 1-3) can have conversion to delirium (ICDSC >/=4).
Mortality | 28 days
  defined as number of days that patients survived in 28 days
Ventilation free days | 28 days
  defined has the number of days from day 1 to day 28 on which a patient breathed without assistance

SECONDARY OUTCOMES:
ICU length of stay | 24 months
  days until ICU discharge
Hospital length of stay | 24 months
  days until ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Paulino, MD, Study Director — Centro Hospitalar de Lisboa Ocidental
Locations (1):
- Maria Carolina Vieira Júlio Paulino, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boettger S, Nunez DG, Meyer R, Richter A, Schubert M, Jenewein J. Subsyndromal delirium in the intensive care setting: Phenomenological characteristics and discrimination of subsyndromal delirium versus no and full-syndromal delirium. Palliat Support Care. 2018 Feb;16(1):3-13. doi: 10.1017/S1478951517000104. Epub 2017 Mar 6. PMID 28262089
- [Background] Brummel NE, Boehm LM, Girard TD, Pandharipande PP, Jackson JC, Hughes CG, Patel MB, Han JH, Vasilevskis EE, Thompson JL, Chandrasekhar R, Bernard GR, Dittus RS, Ely EW. Subsyndromal Delirium and Institutionalization Among Patients With Critical Illness. Am J Crit Care. 2017 Nov;26(6):447-455. doi: 10.4037/ajcc2017263. PMID 29092867
- [Background] Serafim RB, Soares M, Bozza FA, Lapa E Silva JR, Dal-Pizzol F, Paulino MC, Povoa P, Salluh JIF. Outcomes of subsyndromal delirium in ICU: a systematic review and meta-analysis. Crit Care. 2017 Jul 12;21(1):179. doi: 10.1186/s13054-017-1765-3. PMID 28697802
- [Background] Yamada C, Iwawaki Y, Harada K, Fukui M, Morimoto M, Yamanaka R. Frequency and risk factors for subsyndromal delirium in an intensive care unit. Intensive Crit Care Nurs. 2018 Aug;47:15-22. doi: 10.1016/j.iccn.2018.02.010. Epub 2018 Mar 30. PMID 29606481
- [Background] Corona A, Colombo R, Catena E. Early Identification of Subsyndromal Delirium in the Critically Ill: Don't Let the Delirium Rise! Crit Care Med. 2016 Mar;44(3):644-5. doi: 10.1097/CCM.0000000000001544. No abstract available. PMID 26901554